CLINICAL TRIAL: NCT03757546
Title: Extra-pulmonary Clinical Manifestations of Influenza Virus and Respiratory Syncitial Virus Infections
Acronym: GIVRE
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GIVRE
Record Dates: First submitted 2018-10-17; First posted 2018-11-29 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Influenza; Respiratory Virus Syncitial; Extra-respiratory
MeSH Terms: conditions — Influenza, Human | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational — The aim of the study is to describe extra-pulmonary complications due to influenza virus and RSV in hospitalized patients from November 2018 to April 2019 and November 2019 to April 2020 in a French university hospital.

SUMMARY:
The purpose of this study is to describe extra-pulmonary clinical manifestations of Influenza virus and Respiratory Syncitial Virus infections in hospitalized adults at a French university hospital.

DETAILED DESCRIPTION:
Influenza virus and Respiratory Syncitial Virus (RSV) could be responsible for severe infections. Although flu was primarily considered as limited to the respiratory system, clinical reports suggest its association with organ involvement outside of the respiratory tract.

The aim of the study is to describe extra-pulmonary complications due to influenza virus and RSV in hospitalized patients from November 2018 to April 2019 and November 2019 to April 2020 in a French university hospital.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adults ≥18 years old
* Flu or RSV infection confirmed by multiplex qPCR on nasal swab
* Oral non-opposition

Exclusion Criteria:

* No health insurance
* Co-infection with viruses other than influenza or RSV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults hospitalized with flu or RSV infections
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Evaluation frequency of extra-respiratory manifestations with clinical, biological and radiological data | at 1 month
  * Clinical data (clinical examination)
  * Biological Data (blood test)
  * Radiological data

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France